CLINICAL TRIAL: NCT01082380
Title: A Phase One Open-Label Single-Radiolabeled Dose Study To Investigate The Absorption, Metabolism And Excretion Of [14C]PF-02341066 In Healthy Male Volunteers
Brief Title: Radiolabeled [14C]PF-02341066 Study To Investigate The Absorption, Metabolism And Excretion In Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A8081009
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-02

CONDITIONS: Healthy Volunteer
Keywords: radiolabeled; healthy volunteers
MeSH Terms: interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PF-02341066

INTERVENTIONS:
Drug: PF-02341066 — oral suspension, single 250 mg dose of PF 02341066 containing approximately 100 µCi of [14C]PF 02341066
  Other Names: crizotinib

SUMMARY:
The rationale for this study is to investigate the absorption, metabolism and excretion of [14C]PF 02341066 and characterize plasma, fecal and urinary radioactivity, and identify any metabolites, if possible, of [14C]PF 02341066 in humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m^2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081009&StudyName=Radiolabeled%20%5B14C%5DPF-02341066%20Study%20To%20Investigate%20The%20Absorption%2C%20Metabolism%20And%20Excretion%20In%20Healthy%20Male%20Volunteers%20

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-02341066 250 mg: Single oral dose of PF-02341066 250 milligram (mg) containing 100 micro-curie (μCi) Carbon -14[14C].
Period: Overall Study
Arm/Group | PF-02341066 250 mg
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- PF-02341066 250 mg: Single oral dose of PF-02341066 250 mg containing 100 μCi [14C].
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 43.2 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hours (hrs), 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: The Pharmacokinetic (PK) parameter analysis population included all treated participants who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
ng/mL | 109.400 (54.153)

2. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: The PK parameter analysis population included all treated participants who had at least 1 of the PK parameters of primary interest.
Measure: Median (Full Range); unit: hr
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
hr | 2.99 [1.98 to 6.00]

3. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Plasma Concentration (AUClast)
Description: Area under the concentration time-curve from zero to the last measured plasma concentration (AUClast).
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
ng*hr/mL | 2686.0 (1119.6)

4. Primary Outcome: Area Under the Plasma Concentration Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
ng*hr/mL | 2777.0 (1114.9)

5. Primary Outcome: Plasma Decay Half Life (t1/2)
Description: Plasma Decay half-life is the time measured for the concentration to decrease by one half.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
hr | 93.970 (13.797)

6. Primary Outcome: Apparent Oral Clearance (CL/F) of Plasma PF-02341066
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L/hr
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
L/hr | 90.140 (23.984)

7. Primary Outcome: Apparent Volume of Distribution (V/F) in Plasma
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Apparent volume of distribution after oral dose (V/F) is influenced by the fraction absorbed.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
L | 12110.0 (4544.5)

8. Primary Outcome: Renal Clearance (CLr) of PF-02341066
Description: CLr is the volume of plasma from which a substance is completely removed by the kidney in a given amount of time.
Time Frame: Predose, 0 to 4, 4 to 8, 8 to 16, 16 to 24 to 36, 36 to 48 hrs and then after every 24 hrs until up to 480 hrs post-dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L/hr
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
L/hr | 2.11 (0.29)

9. Primary Outcome: Total Amount of Unchanged Drug Excreted in the Urine From Time Zero to Infinite Time (Ae)
Description: Ae = concentration of unchanged drug excreted in the urine multiplied by volume of unchanged drug excreted in urine.
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: mg
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
mg | 5.847 (3.450)

10. Primary Outcome: Total Amount of Unchanged Drug Excreted in the Urine Expressed as Percent of Dose From Time Zero to Infinite Time [Ae(%)]
Time Frame: as for outcome 8
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Percent dose of unchanged drug
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
Percent dose of unchanged drug | 2.339 (1.380)

11. Primary Outcome: Maximum Observed Concentration in Plasma Radioactivity (Cmax)
Description: Radioactivity corresponds to 100 μCi [14C]PF-02341066.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: The radioactivity parameter analysis population included all treated participants who had at least 1 of the radioactivity parameters of primary interest.
Measure: Geometric Mean (Standard Deviation); unit: nanogram-equivalent/milliliter(ng-eq/mL)
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
nanogram-equivalent/milliliter(ng-eq/mL) | 435.600 (82.072)

12. Primary Outcome: Time to Reach Maximum Observed Plasma Radioactivity Concentration (Tmax)
Description: Radioactivity corresponds to 100 μCi [14C]PF-02341066.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: as for outcome 11
Measure: Median (Full Range); unit: hr
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
hr | 5.00 [2.98 to 6.00]

13. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Plasma Radioactivity Concentration (AUClast)
Description: Area under the concentration time-curve from zero to the last measured plasma concentration. Radioactivity corresponds to 100 μCi [14C]PF-02341066.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: ng-eq*hr/mL
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
ng-eq*hr/mL | 22830.0 (2636.4)

14. Primary Outcome: Area Under the Plasma Radioactivity Concentration Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Description: Area under the concentration curve from time zero to extrapolated infinite time [AUC (0 - ∞)] in plasma. Radioactivity corresponds to 100 μCi [14C]PF-02341066.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: Data was insufficient to analyze as only 2 participants were evaluable for the parameter.
Measure: Geometric Mean (Standard Deviation); unit: ng-eq*hr/mL
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 0

15. Primary Outcome: Decay Half Life (t1/2) of Radioactivity in Plasma
Description: Plasma decay half-life is the time measured for the plasma radioactivity concentration to decrease by one half. Radioactivity corresponds to 100 μCi [14C]PF-02341066.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: Data was insufficient to analyze as only 2 participants were evaluable for the parameter.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 0

16. Primary Outcome: Apparent Oral Clearance (CL/F) of Plasma Radioactivity
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Radioactivity corresponds to 100 μCi [14C]PF-02341066.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: Data was insufficient to analyze as only 2 participants were evaluable for the parameter.
Measure: Geometric Mean (Standard Deviation); unit: L/hr
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 0

17. Primary Outcome: Apparent Volume of Distribution (V/F) in Plasma Radioactivity
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Apparent volume of distribution after oral dose (V/F) is influenced by the fraction absorbed. Radioactivity corresponds to 100 μCi [14C]PF-02341066.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: Data was insufficient to analyze as only 2 participants were evaluable for the parameter.
Measure: Geometric Mean (Standard Deviation); unit: L
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 0

18. Primary Outcome: Maximum Observed Concentration of Radioactivity in Whole Blood (Cmax)
Description: Radioactivity corresponds to 100 μCi [14C]PF-02341066.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: ng-eq/mL
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
ng-eq/mL | 312.300 (62.669)

19. Primary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of Radioactivity in Whole Blood
Description: Time to Reach Maximum Observed Concentration (Tmax) of Radioactivity in whole blood. Radioactivity corresponds to 100 μCi [14C]PF-02341066.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: as for outcome 11
Measure: Median (Full Range); unit: hr
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
hr | 4.00 [2.98 to 6.00]

20. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Radioactivity in Whole Blood
Description: Area under the concentration time-curve from zero to the last measured concentration (AUClast) in whole blood. Radioactivity corresponds to 100 μCi [14C]PF-02341066.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: as for outcome 11
Measure: Geometric Mean (Standard Deviation); unit: ng-eq*hr/mL
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
ng-eq*hr/mL | 7032.0 (1284.2)

21. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of Radioactivity in Whole Blood
Description: Area under the concentration curve from time zero to extrapolated infinite time [AUC (0 - ∞)] in whole blood. Radioactivity corresponds to 100 μCi [14C]PF-02341066.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: Data was insufficient to analyze as only 2 participants were evaluable for the parameter.
Measure: Geometric Mean (Standard Deviation); unit: ng-eq*hr/mL
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 0

22. Primary Outcome: Decay Half-life (t1/2) of Radioactivity in Whole Blood
Description: Decay half life (t1/2) is the time measured for the concentration to decrease by one half in whole blood. Radioactivity corresponds to 100 μCi [14C]PF-02341066.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: Data was insufficient to analyze as only 2 participants were evaluable for the parameter.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 0

23. Primary Outcome: Apparent Oral Clearance of Radioactivity From Whole Blood (CL/F)
Description: as for outcome 16
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: Data was insufficient to analyze as only 2 participants were evaluable for the parameter.
Measure: Geometric Mean (Standard Deviation); unit: L/hr
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 0

24. Primary Outcome: Apparent Volume of Distribution of Radioactivity in Whole Blood (V/F)
Description: as for outcome 17
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: Data was insufficient to analyze as only 2 participants were evaluable for the parameter.
Measure: Geometric Mean (Standard Deviation); unit: L
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 0

25. Primary Outcome: Total [14C] Data in Urine
Description: Cumulative amount excreted in urine at specified intervals after administration of a single 250-mg (100 μCi) oral dose of [14C]PF-02341066.
Time Frame: as for outcome 8
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng-eq
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
ng-eq | 56200000 (11500000)

26. Primary Outcome: Total [14C] Data in Feces
Description: Cumulative amount excreted in feces at specified intervals after administration of a single 250-mg (100 μCi) oral dose of [14C]PF-02341066.
Time Frame: From Day 0 through pre-dose (Day1) and as passed through until up to 480 hrs post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng-eq
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
ng-eq | 160000000 (15000000)

27. Primary Outcome: Overall Cumulative Percent Recovery of Radioactivity
Description: Overall cumulative percent of radioactive dose recovered in urine, feces and toilet tissue at specified intervals after administration of a single 250-mg (100 μCi) oral dose of [14C]PF-02341066.
Time Frame: Pre-dose, 0 to 4, 4 to 8, 8 to 16, 16 to 24 to 36, 36 to 48 hrs and then after every 24 hrs until up to 480 hrs post-dose for urine and Day 0 through pre-dose (Day1) and as passed through until up to 480 hrs post-dose for feces
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent recovery of radioactivity
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
Percent recovery of radioactivity
  Urine | 22.20 (4.63)
  Feces | 63.10 (5.93)
  Overall | 85.20 (8.38)

28. Primary Outcome: Identification and Profiling of Metabolites of [14C]PF-02341066 in Plasma
Description: Identification was done by Radio-High Performance liquid chromatography (HPLC) chromatogram. Relative abundance (profiling) of metabolites in chromatogram were determined by dividing sum of radioactive content of fractions contributing to particular peak by sum of radioactive content of all fractions constructing the radio chromatogram. Metabolites accounting for an average of greater than or equal to (>=) 10% of total recoverable radioactivity in plasma were summarized. Radioactivity corresponds to 100 μCi [14C] PF-02341066.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24 hrs, 36 hrs, 48 hrs, then after every 24 hrs until up to 480 hrs post-dose
Population: as for outcome 11
Measure: Number; unit: Percentage of recovered radioactivity
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
Percentage of recovered radioactivity
  PF-02341066 | 33.1
  M10, PF-06260182 | 10.2

29. Primary Outcome: Identification and Profiling of Metabolites of [14C]PF-02341066 in Feces
Description: In feces, metabolite abundance (profiling) was calculated by multiplying the fractional contribution of radioactive response for the peak in the Radio-HPLC chromatogram to the total radioactivity detected by the percent of administered dose recovered in the matrix. Only those metabolites that were a component of a chromatographic peak that accounted for an average of >=1% of the administered dose, were summarized. Radioactivity corresponds to 100 μCi [14C] PF-02341066.
Time Frame: From Day 0 through pre-dose (Day1) and as passed through until up to 480 hrs post-dose
Population: as for outcome 11
Measure: Number; unit: Percentage of radioactive dose
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
Percentage of radioactive dose
  PF-02341066 | 53.5
  M8 | NA — Data was collected but could not be quantified.

30. Primary Outcome: Identification and Profiling of Metabolites of [14C]PF-02341066 in Urine
Description: In urine, metabolite abundance (profiling) was calculated by multiplying the fractional contribution of radioactive response for the peak in the Radio-HPLC chromatogram to the total radioactivity detected by the percent of administered dose recovered in the matrix. Only those metabolites that were a component of a chromatographic peak that accounted for an average of >=1% of the administered dose, were summarized. Radioactivity corresponds to 100 μCi [14C] PF-02341066.
Time Frame: as for outcome 8
Population: as for outcome 11
Measure: Number; unit: Percentage of radioactive dose
Arm/Group | PF-02341066 250 mg
Number analyzed (Participants) | 6
Percentage of radioactive dose
  PF-02341066 | 2.4
  M8 | 4.5

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-02341066 250 mg
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02341066 250 mg (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Somnolence (Nervous system disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes